CLINICAL TRIAL: NCT01382511
Title: Simvastatin Treatment of Pachyonychia Congenita
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Department of Dermatology, Tel Aviv Sourasky Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0462-09-TLV
Record Dates: First submitted 2011-06-14; First posted 2011-06-27 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2009-10

CONDITIONS: Pachyonychia Congenita
MeSH Terms: conditions — Pachyonychia Congenita | interventions — Simvastatin

INTERVENTIONS:
Drug: Simvastatine — 80 mg

SUMMARY:
Simvastatin and related statins, such as compactin, are able to inhibit the constitutive expression of inducible/repressible keratin genes such as K6a and K17. This effect is due to the reported ability of statins to inhibit STAT1 expression (Lee et al., 2007). The constitutive K6a promoter activity is dependent on STAT1 and blocked by simvastatin or siRNA against STAT1. This STAT1-dependent constitutive expression of K6a, is independent of JAK (Janus family of kinases).

Thus simvastatin is capable of down-regulating both the constitutive and interferon-inducible expression of PC-related keratins such as K6a and K17. Therefore, this class of molecule has potential for the treatment of PC or related inherited disorders where the causative mutation resides in an inducible/repressible keratin gene such as K6a or K17.

Simvastatin or other statins approved for human use might be delivered either orally, as is currently the case for cholesterol-lowering treatment or, if higher therapeutic doses are required in skin for reduction of hyperkeratosis in PC or in related keratinizing disorders, this might be achieved by topical formulations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pachyonychia congenita with known mutations in keratin 6a. -

Exclusion Criteria:

* The use of concomitant medications known to interact with simvastatin.
* This would include itraconazole, ketoconazole, fluconazole, gemfibrozil, verapamil, diltiazem, mibefradil, erythromycin, clarithromycin, telithromycin, cyclosporine, ritonavir, nefazodone, danazol, amiodarone, Rifampin, and carbamazepine.
* During the study subjects must agree to avoid grapefruit juice.
* Also excluded are patients with a past history of myopathy, or impaired liver function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2011-07; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of decreased hyperkeratosis | six months
  Decreased hyperkeratosis